CLINICAL TRIAL: NCT00380133
Title: A Randomised, Double-blind, Double-dummy, Placebo-controlled, Five-way Crossover Study to Assess the Effects of Single Oral Doses of SB-681323 (7.5 mg and 25 mg) and Prednisolone (10 mg and 30 mg) on Biomarkers in Induced Sputum and Blood in COPD Patients.
Brief Title: Study of SB681323 and Prednisolone on Biomarkers in COPD (Chronic Obstructive Pulmonary Disease) Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IPI100477
Record Dates: First submitted 2006-09-21; First posted 2006-09-25 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2012-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD SB-681323 prednisolone biomarkers
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — dilmapimod; Prednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (1):
- Randomised, double-blind, five-way crossover (Experimental): A randomised, double-blind, double-dummy, placebo-controlled, five-way crossover study to assess the effects of single oral doses of SB-681323 (7.5 mg and 25 mg) and prednisolone (10 mg and 30 mg) on biomarkers in induced sputum and blood in COPD patients.
  Interventions: Drug: SB681323; Drug: Prednisolone; Drug: Placebo

INTERVENTIONS:
Drug: SB681323 — 5 mg and 2.5 mg tablets - The tablets will be round (9.0 mm in diameter) and white and provided in labelled bottles
Drug: Prednisolone — 5 mg size DB AA capsule shell (Swedish orange) with a powder backfill (lactose Anhydrous)
Drug: Placebo — Tablets matched to SB681323 or prednisolone

SUMMARY:
This study will assess the effects of single oral doses of SB681323 and prednisolone on biomarkers in induced sputum and blood COPD patients

ELIGIBILITY:
Inclusion criteria:

* Subject is current smoker or ex-smoker with a smoking history of at least 10 pack years (number of pack years = [number of cigarettes per day/20] x number of years smoked).
* The patient has serum CRP ≥ 3 mg/L at screening
* Subjects able to understand and comply with protocol requirements, instructions and protocol-stated restrictions.

Exclusion criteria:

* Any clinically relevant abnormality identified on medical assessment, laboratory examination, or 12-lead ECG which in the opinion of the investigator, will lead to an unacceptable increase in the risk of study participation or will call into question the validity of the outcome measures.
* Subjects who are obese, defined as having a BMI > 40
* Subject has a diagnosis of asthma that is confirmed by the investigator.
* Subject has poorly controlled COPD, defined as the occurrence of any of the following in the 2 weeks prior to visit 1: acute worsening of COPD that is managed by the subject at home by self-treatment with corticosteroids or antibiotics, or that requires treatment by a physician.
* Subject has active tuberculosis, lung cancer or clinically overt bronchiectasis.
* Symptoms of "cold or flu" or any respiratory infection/symptoms at the start of the study
* Subject has cardiac, gastrointestinal, neurological, renal, endocrine or psychiatric disease that is uncontrolled on permitted medication
* Subject has history of allergic rhinitis.
* Subjects with a history of any type of malignancy with the exception of successfully treated basal cell cancer of the skin.
* Subjects with rheumatoid arthritis, connective tissue disorders and other conditions known to be associated with chronic inflammation (e.g. Inflammatory Bowel Disease).
* Subjects with chronic infections such as gingivitis, periodontitis, prostatitis, gastritis, and urinary tract infections.
* Subjects with history of hepatic disease.
* History of increased liver function tests (ALT, AST) above upper limit of normal in the past 6 months and/or liver function tests (bilirubin, ALT, AST) above upper limit of normal at screening.
* History of positive HIV, Hepatitis B /C antibody test result, a positive Hep B/C result at screen or a risk factor for these diseases.
* History of drug or other allergy, which, in the opinion of the Investigator precludes participation in the study.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-06; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamic effect of single, oral doses of SB-681323 and prednisolone | 20 weeks
  Levels of ex-vivo LPS induced TNFα in whole blood at 1, 2, 6 and 24 hrs post-dose

SECONDARY OUTCOMES:
Level of pHSP27 and mRNAs encoding inflammatory markers | 20 weeks
  Levels obtained in sputum and whole blood samples
CD11b and CD62L surface expression on neutrophils | 20 weeks
  Levels obtained in whole blood samples
Blood concentration of inflammatory markers | 20 weeks
  GSK's COPD multiplex biomarker assay
CRP levels | 20 weeks
  Levels obtained in COPD patient sera
Safety and tolerability of dinsgle doses of SB681323 and prednisolone | 20 weeks
  Vitals, AEs, ECGs, safety laboratory, pulmonary function FEV1 and FVC
Exploratory objective #1 | 20 weeks
  Transcriptomic profiles of induced sputum cells and whole blood Exploratory micro-array analysis of mRNA biomarkers in induced sputum samples at 2 hrs post-dose and whole blood samples at baseline (pre-dose), and 6 hrs post-dose (earlier post-dose blood samples (1 and 2 hrs ) may also be examined)
Exploratory objective #2 | 20 weeks
  Exploratory analysis of inflammatory biomarker concentrations in induced sputum supernatants (e.g. myeloperoxidase, IL-6, TNF-α, total protein) at 2 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Manchester, Lancashire, United Kingdom

REFERENCES:
- [Derived] Singh D, Smyth L, Borrill Z, Sweeney L, Tal-Singer R. A randomized, placebo-controlled study of the effects of the p38 MAPK inhibitor SB-681323 on blood biomarkers of inflammation in COPD patients. J Clin Pharmacol. 2010 Jan;50(1):94-100. doi: 10.1177/0091270009347873. Epub 2009 Oct 30. PMID 19880675